CLINICAL TRIAL: NCT04728230
Title: A Phase I/II Trial of PARP Inhibition, Radiation, and Immunotherapy in Patients With Extensive-Stage Small Cell Lung Cancer (ES-SCLC) - PRIO Trial
Brief Title: Olaparib and Durvalumab With Carboplatin, Etoposide, and/or Radiation Therapy for the Treatment of Extensive-Stage Small Cell Lung Cancer, PRIO Trial
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0612; NCI-2020-06178 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0612 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-31; First posted 2021-01-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; durvalumab; Immunoglobulin G; Disulfides; Etoposide; olaparib; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemo-immunotherapy, radiation therapy) (Experimental): See detailed description.
  Interventions: Drug: Carboplatin; Biological: Durvalumab; Drug: Etoposide; Drug: Olaparib; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
Radiation: Radiation Therapy — Undergo consolidative thoracic radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I/II trials investigates the side effects of olaparib and durvalumab and how well it works in combination with carboplatin, etoposide, and/or radiation therapy in treating patients with extensive stage-small cell lung cancer (ES-SCLC) who have not received treatment for their disease. PARPs are proteins that help repair DNA mutations. PARP inhibitors, such as olaparib, can keep PARP from working, so tumor cells can't repair themselves, and they may stop growing. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as carboplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy sources to kill tumor cells and shrink tumors. Giving olaparib and durvalumab together with carboplatin, etoposide, and/or radiation therapy may help treat patients with ES-SCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the toxicity and feasibility of sequential treatment with olaparib, thoracic radiotherapy (TRT)/durvalumab, and olaparib/durvalumab for consolidation and maintenance therapy in patients status post (s/p) chemoimmunotherapy for ES-SCLC.

SECONDARY OBJECTIVE:

I. To assess the efficacy of sequential treatment with olaparib, TRT/durvalumab, and olaparib/durvalumab for consolidation and maintenance therapy in patients s/p chemoimmunotherapy for ES-SCLC.

EXPLORATORY OBJECTIVES:

I. Perform a comparative analysis of patient clinical outcome according to tumor biomarkers in circulating tumor cell (CTC), blood samples and tumor tissue, such as SLFN11 expression H- scores and stratifying tumors as SLFN11 positive or negative on the basis of H-score >= 1.

II. Perform a comparative analysis of patient clinical outcome according to immune biomarkers in blood and tumor tissue, such as PD-L1 immunohistochemistry (IHC) 22C3 pharmDx assay and stratifying tumors as PD-L1 positive or negative on the basis of PD-L1 combined positive score >= 1% in patients treated with anti- PD-L1 therapy.

III. Perform whole exome sequencing (WES) and methylation profiling on tumor samples and from circulating-free deoxyribonucleic acid (cfDNA) to evaluate whether tumor mutational burden (TMB) or specific genomic alterations are associated with improved progression free survival (PFS) with the trial regimen.

IV. Gene and protein expression of tumor tissue through ribonucleic acid (RNA) sequencing and Reverse Phase Protein Array (RPPA).

V. Quantify pre-treatment, pre- and post-olaparib, post-TRT, and at progression levels for blood-based biomarkers, such as cytokines associated with immune activation (e.g., STING pathway cytokines, CXCL10 and CCL5) to establish correlations with PFS and overall survival (OS).

VI. Using longitudinal blood samples (e.g. pre-treatment, pre- and post-olaparib, post-TRT, and at progression), assess CTC number, CTC (single-cell) biomarker expression (such as SLFN11 and PD-L1 expression), and immune profile of PBMCs.

VIa. Correlate baseline expression or changes with PFS and OS. VII. Assess pre- and post-olaparib, and at progression tumor tissue for immune markers, such as CD8+ T cells, through multiplex IHC.

VIII. Assessment of single-cell biomarker expression on CTCs and tumor tissue (such as SLFN11 and PD-L1 expression) and immune profile of peripheral blood mononuclear cells (PBMCs).

VIIIa. Correlate pre-treatment expression or changes with PFS and/or OS. IX. Generation of CTC-derived and/or biopsy-derived xenograft models from individual patients

OUTLINE:

CHEMO-IMMUNOTHERAPY: Patients receive durvalumab intravenously (IV) over 60 minutes on day 1, carboplatin IV over 60 minutes on day 1, etoposide IV over 60 minutes on days 1-3. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with response or stable disease (SD) after cycle 4 and are candidates for TRT proceed to Induction. Patients that are not candidates for TRT proceed to Single-Agent Maintenance.

INDUCTION (WEEKS 13-14): Patients receive olaparib orally (PO) twice daily (BID) on days 1-11 in the absence of disease progression or unacceptable toxicity.

IMMUNORADIATION (WEEKS 15-18): Patients receive durvalumab IV over 60 minutes on day 1. Patients also undergo consolidative TRT daily on days 1-5 and 8-12 in the absence of disease progression or unacceptable toxicity.

MAINTENANCE (WEEKS 19 AND BEYOND): Patients without progressive disease receive durvalumab IV over 60 minutes on day 1, and olaparib PO BID. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

SINGLE-AGENT MAINTENANCE: Patients receive durvalumab IV over 60 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 30 days, then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written informed consent form prior to any mandatory study specific procedures, sampling, and analyses. For inclusion in i) the optional exploratory genetic research and ii) the optional biomarker research, patients must fulfill the following criteria:

  * Provision of informed consent for genetic research prior to collection of sample;
  * Provision of informed consent for biomarker research prior to collection of sample;
  * If a patient declines to participate in the optional exploratory genetic research or the optional biomarker research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by computed tomography (CT) and is suitable for repeated assessment
* Patients with previously treated brain metastases that are asymptomatic for at least 14 days and only require prednisone equivalent of 10 mg daily or less prior to study treatment
* Histological or cytological documented ES-SCLC: American Joint Committee on Cancer (AJCC) stage IV SCLC (T any, N any, M1 a/b), including patients with T3-4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan
* No prior systemic therapy for ES-SCLC, including, but not limited to, chemotherapy, PARP inhibitor, and PD-1/PD-L1 checkpoint inhibitors. Palliative radiation is allowed if completed a minimum of three days prior to beginning of study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 at enrollment
* Body weight > 30 kg
* Hemoglobin >=10.0 g/dL with no blood transfusion in the past 28 days (measured within 28 days prior to administration of study treatment)
* Absolute neutrophil count >= 1.5 x 10^9 /L (measured within 28 days prior to administration of study treatment)
* Platelet count >= 100 x 10^9/L (measured within 28 days prior to administration of study treatment)
* Serum bilirubin =<1.5 x institutional upper limit of normal (ULN) (measured within 28 days prior to administration of study treatment)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x institutional ULN, unless liver metastases are present in which case they must be =< 5 x ULN (measured within 28 days prior to administration of study treatment)
* Calculated estimated creatinine clearance >= 51 mL/min using the Cockcroft- Gault equation or based on a 24-hour urine test (measured within 28 days prior to administration of study treatment)
* Evidence of post-menopausal status or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1. Postmenopausal status is defined as:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50
  * Radiation-induced oophorectomy with last menses > 1 year ago
  * Chemotherapy-induced menopause with > 1-year interval since last menses
  * Surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women of childbearing potential and their partners, who are sexually active, must agree to the use of TWO highly effective forms of contraception in combination. This should be started from the signing of the informed consent and continue throughout the period of taking study treatment and for at least 3 months after last dose of study drug(s)
  * Male patients must use a condom during treatment and for 3 months after the last dose of study treatment when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential. Male patients should not donate sperm throughout the period of taking study treatment and for 3 months following the last dose of study treatment
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up

Exclusion Criteria:

* Histology other than SCLC
* Prior systemic therapy for ES-SCLC (e.g. chemotherapy, PARP inhibitor, other DNA damage response [DDR] inhibitors, PD-1/PD-L1 inhibitors)
* Patients with untreated brain metastases
* Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study treatment and patients must have recovered from any effects of any major surgery. Note: Local surgery of isolated lesions for palliative intent is acceptable
* Other malignancy unless curatively treated with no evidence of disease for >= 3 years except:

  * Adequately treated non-melanoma skin cancer.
  * Curatively treated in situ cancer of the cervix; ductal carcinoma in situ (DCIS); stage 1, grade 1 endometrial carcinoma; and in situ bladder cancer
* Any concurrent anticancer therapy
* Resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g. unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QT corrected by Fridericia [QTcF] prolongation > 500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome
* Current or prior use of immunosuppressive medication within 14 days prior to cycle 1 (C1) of study treatment, with the exceptions of intranasal and inhaled corticosteroids, or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone or an equivalent corticosteroid
* Active or prior documented autoimmune disease within the past 2 years. NOTE: vitiligo, alopecia, chronic skin condition that does not require systemic therapy, psoriasis not requiring systemic treatment (within the past 2 years), and hypothyroidism (if stable on hormonal therapy) are not exclusion criteria
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis) or pneumonitis
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV)
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Patients considered high medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent
* Patients with myelodysplastic syndrome (MDS) / acute myeloid leukemia (AML) or with features suggestive of MDS/AML
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable outside of 28 days prior to treatment)
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks
* Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
* Participation in another clinical study with an investigational product (IP) administered in the last 6 months
* Involvement in the planning and/or conduct of the study
* Previous enrollment in the present study
* Receipt of live attenuated vaccination within 30 days prior to study entry
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing two highly effective methods of birth control
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Known allergy or hypersensitivity to durvalumab, olaparib or any excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity | From start of olaparib, at the end of cycle 6 (each cycle is 28 days)
  Will be assessed per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Toxicity data by type and severity will be summarized in frequency tables.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Time from starting chemo-immunotherapy until disease progression or death from any cause, assessed up to 1 year
  Assessed per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. PFS will be compared to the pre-specified parameter obtained from historical data of comparable patients with extensive-stage small cell lung cancer (ES-SCLC) treated with frontline etoposide plus either cisplatin or carboplatin (EP) chemotherapy followed by thoracic radiation. Will be estimated using the Kaplan-Meier method. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Cox regression model will be applied to evaluate the effect of potential covariates on PFS.
Overall survival (OS) | Time from starting chemo-immunotherapy until death from any cause, assessed up to 1 year
  Will be estimated using the Kaplan-Meier method. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Cox regression model will be applied to evaluate the effect of potential covariates on OS.
Overall response rate (ORR) | Up to 1 year
  The patient's best overall response assignment will depend on the findings of both target and non-target disease and will also take into consideration the appearance of new lesions.
Intra- and extra-thoracic recurrence rates | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo V Negrao, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org